CLINICAL TRIAL: NCT05028231
Title: Neoadjuvant Immunotherapy (PD-1 / PD-L1) Combined With Chemotherapy for Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma: a Single Center, Prospective, Open, One Arm Exploratory Clinical Study
Acronym: NICCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Zhang Ni, Proffesor, Tongji Hospital
Other Study IDs: TJ-IRB20210624
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Esophageal Squamous Cell Carcinoma; Neoadjuvant Therapies
Keywords: Immunotherapy; Chemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue samples will be taken before and after treatment for gene testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Neoadjuvant Immunotherapy (PD-1 / PD-L1) Combined With Chemotherapy
  Interventions: Procedure: Neoadjuvant Immunotherapy (PD-1 / PD-L1) Combined With Chemotherapy

INTERVENTIONS:
Procedure: Neoadjuvant Immunotherapy (PD-1 / PD-L1) Combined With Chemotherapy — Each patient will complete 2 cycles of neoadjuvant therapy. After evaluating the curative effect, decide whether to operate or not. Patients with and without surgery enter the survival follow-up period.

SUMMARY:
To purpose of this study is to access the safety and efficacy of neoadjuvant Immunotherapy (PD-1 / PD-L1) combined with chemotherapy for locally advanced thoracic esophageal squamous cellcarcinoma.

DETAILED DESCRIPTION:
Each patient will complete 2 cycles of neoadjuvant therapy and decide whether to operate after evaluating the curative effect if there is no active withdrawal of the subject from the trial or the researcher believes that the subject is not suitable for further trials. The patients after operation and without operation enter the survival follow-up period. If the imaging evaluation is PD after neoadjuvant therapy, the follow-up treatment shall be carried out according to the following principles: the imaging evaluation belongs to the continuous operation that can be operated; If the imaging evaluation was inoperable, radical concurrent radiotherapy and chemotherapy were performed. Postoperative adjuvant therapy shall be performed according to NCCN guidelines. If it is necessary to improve the local control rate, postoperative adjuvant radiotherapy is feasible. At the same time, imaging evaluation was performed until tumor recurrence and metastasis. After tumor recurrence and metastasis, all patients should also enter survival follow-up; In case of drug withdrawal (such as intolerable toxicity) other than recurrence and metastasis during treatment, the treatment is completed, the post-treatment visit is entered, and the survival follow-up is entered after recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 Years old，
* The clinical stage of esophageal cancer confirmed by pathology was cT（1-3）N（1-3）M0
* No previous chemoradiotherapy
* ECOG PS: 0-1 points
* The functions of important organs meet the following requirements (excluding the use of any blood components and cell growth factors during the screening period)：Absolute neutrophil count ≥ 1.5 × 109/L； Platelet ≥ 90 × 109/L； Hemoglobin ≥ 9g / dl; Serum albumin ≥ 3G / dl; Thyroid stimulating hormone (TSH) ≤ ULN (if abnormal, the levels of T3 and T4 should be investigated at the same time. If the levels of T3 and T4 are normal, they can be included in the group); Bilirubin ≤ ULN; ALT and AST ≤ 1.5 times ULN; AKP ≤ 2.5 times ULN; Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60ml / min.
* Women of childbearing age must have taken reliable contraceptive measures or conducted pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and are willing to use appropriate contraceptive methods during the test and 8 weeks after the last administration of test drugs. For men, they must agree to use appropriate methods of contraception or surgical sterilization during the trial and 8 weeks after the last administration of the trial drug.
* The patients voluntarily joined the study and signed the informed consent form. They had good compliance and cooperated with the follow-up.

Exclusion Criteria:

* Any active autoimmune disease or history of autoimmunity (as follows, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism and hypothyroidism; Subjects with vitiligo or asthma in childhood have been completely relieved and do not need any intervention after adulthood can be included; Asthma in which subjects need bronchodilators for medical intervention cannot be included).
* Those who have used other drugs in clinical trials within 4 weeks before the first medication.
* Severe allergic reaction to monoclonal antibody.
* The number of neutrophils in peripheral blood was less than 1500 / mm3.
* There are cardiac clinical symptoms or diseases that are not well controlled.
* Previously received radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeted therapy.
* The subjects were innate or acquired immunodeficiency (such as HIV), or active hepatitis (hepatitis B reference: HBsAg) positive, HBVDNA > 2000IU/ml or copy number > 104/ml; Hepatitis C reference: HCV antibody positive.
* According to the judgment of the researcher, the subject has other factors that may lead to the forced midway termination of this study, such as other serious diseases (including mental diseases) requiring combined treatment, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subject, or the collection of data and samples.
* The researchers judged the patients with high risk of esophageal perforation or no potential possibility of surgery through endoscopic ultrasonography or imaging.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this clinical trial, patients with resectable thoracic esophageal squamous cell carcinoma can receive neoadjuvant immunotherapy and neoadjuvant chemotherapy before operation.
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | 2-5 years
  According to the detection of pathological specimens after operation, no malignant tumor cells were detected, so the patient achieved complete pathological remission.

SECONDARY OUTCOMES:
Disease-free Survival | 2-5 years
  The patient achieved CR (complete remission) and still had no probability of recurrence after treatment in 2-years.
Progression-Free-Survival | 2-5 years
  The time between the beginning of treatment and the observation of disease progression or death from any cause.
Overall survival | 2-5 years
  The time from randomization to death from any cause.
Security | 2-5 years
  The safety of drugs was evaluated from four aspects: adverse events, adverse reactions, serious adverse events and serious adverse reactions.
Objective Response Rate | 2-5 years
  The proportion of patients whose tumor volume reduced to a predetermined value and could maintain the minimum time limit.

OTHER OUTCOMES:
Tumor markers | 2-5 years
  Tumor markers refer to those characteristic bioactive substances that can be detected that can reflect the development stage of malignant tumor cells. In a narrow sense, tumor markers refer to bioactive substances synthesized, secreted and released into blood and / or body fluid by malignant tumor cells, including enzymes, hormones, proteins, metabolites and other substances, Their occurrence and changes are closely related to the growth, diffusion, occurrence and development of malignant tumors.
Intestinal flora | 2-5 years
  Intestinal flora homeostasis is called the organ of human body. Intestinal flora homeostasis plays an important role in the life activities of the body. It has important physiological significance in promoting the digestion and absorption of host nutrients, maintaining the normal physiological function of intestine, regulating body immunity and antagonizing the colonization of pathogenic microorganisms.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Wuhan, Hubei Provience, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pennathur A, Gibson MK, Jobe BA, Luketich JD. Oesophageal carcinoma. Lancet. 2013 Feb 2;381(9864):400-12. doi: 10.1016/S0140-6736(12)60643-6. PMID 23374478
- [Background] Chen MF, Chen PT, Chen WC, Lu MS, Lin PY, Lee KD. The role of PD-L1 in the radiation response and prognosis for esophageal squamous cell carcinoma related to IL-6 and T-cell immunosuppression. Oncotarget. 2016 Feb 16;7(7):7913-24. doi: 10.18632/oncotarget.6861. PMID 26761210
- [Background] Chen K, Cheng G, Zhang F, Zhang N, Li D, Jin J, Wu J, Ying L, Mao W, Su D. Prognostic significance of programmed death-1 and programmed death-ligand 1 expression in patients with esophageal squamous cell carcinoma. Oncotarget. 2016 May 24;7(21):30772-80. doi: 10.18632/oncotarget.8956. PMID 27120796
- [Result] Sjoquist KM, Burmeister BH, Smithers BM, Zalcberg JR, Simes RJ, Barbour A, Gebski V; Australasian Gastro-Intestinal Trials Group. Survival after neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal carcinoma: an updated meta-analysis. Lancet Oncol. 2011 Jul;12(7):681-92. doi: 10.1016/S1470-2045(11)70142-5. Epub 2011 Jun 16. PMID 21684205
- [Result] Apinop C, Puttisak P, Preecha N. A prospective study of combined therapy in esophageal cancer. Hepatogastroenterology. 1994 Aug;41(4):391-3. PMID 7959579
- [Result] Walsh TN, Noonan N, Hollywood D, Kelly A, Keeling N, Hennessy TP. A comparison of multimodal therapy and surgery for esophageal adenocarcinoma. N Engl J Med. 1996 Aug 15;335(7):462-7. doi: 10.1056/NEJM199608153350702. PMID 8672151
- [Result] Urba SG, Orringer MB, Turrisi A, Iannettoni M, Forastiere A, Strawderman M. Randomized trial of preoperative chemoradiation versus surgery alone in patients with locoregional esophageal carcinoma. J Clin Oncol. 2001 Jan 15;19(2):305-13. doi: 10.1200/JCO.2001.19.2.305. PMID 11208820
- [Result] Lee JL, Park SI, Kim SB, Jung HY, Lee GH, Kim JH, Song HY, Cho KJ, Kim WK, Lee JS, Kim SH, Min YI. A single institutional phase III trial of preoperative chemotherapy with hyperfractionation radiotherapy plus surgery versus surgery alone for resectable esophageal squamous cell carcinoma. Ann Oncol. 2004 Jun;15(6):947-54. doi: 10.1093/annonc/mdh219. PMID 15151953
- [Result] Burmeister BH, Smithers BM, Gebski V, Fitzgerald L, Simes RJ, Devitt P, Ackland S, Gotley DC, Joseph D, Millar J, North J, Walpole ET, Denham JW; Trans-Tasman Radiation Oncology Group; Australasian Gastro-Intestinal Trials Group. Surgery alone versus chemoradiotherapy followed by surgery for resectable cancer of the oesophagus: a randomised controlled phase III trial. Lancet Oncol. 2005 Sep;6(9):659-68. doi: 10.1016/S1470-2045(05)70288-6. PMID 16129366
- [Result] Tepper J, Krasna MJ, Niedzwiecki D, Hollis D, Reed CE, Goldberg R, Kiel K, Willett C, Sugarbaker D, Mayer R. Phase III trial of trimodality therapy with cisplatin, fluorouracil, radiotherapy, and surgery compared with surgery alone for esophageal cancer: CALGB 9781. J Clin Oncol. 2008 Mar 1;26(7):1086-92. doi: 10.1200/JCO.2007.12.9593. PMID 18309943
- [Result] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] Lim SH, Hong M, Ahn S, Choi YL, Kim KM, Oh D, Ahn YC, Jung SH, Ahn MJ, Park K, Zo JI, Shim YM, Sun JM. Changes in tumour expression of programmed death-ligand 1 after neoadjuvant concurrent chemoradiotherapy in patients with squamous oesophageal cancer. Eur J Cancer. 2016 Jan;52:1-9. doi: 10.1016/j.ejca.2015.09.019. Epub 2015 Nov 26. PMID 26623522
- [Result] Huang J, Xu B, Mo H, Zhang W, Chen X, Wu D, Qu D, Wang X, Lan B, Yang B, Wang P, Zhang H, Yang Q, Jiao Y. Safety, Activity, and Biomarkers of SHR-1210, an Anti-PD-1 Antibody, for Patients with Advanced Esophageal Carcinoma. Clin Cancer Res. 2018 Mar 15;24(6):1296-1304. doi: 10.1158/1078-0432.CCR-17-2439. Epub 2018 Jan 22. PMID 29358502
- [Derived] Deng S, Wang Q, Li Y, Zhang R, Li J, Zhang Y, Cai Y, Sun W, Chang J, Zhang N, Zhang L. Clinical efficacy and biomarkers of neoadjuvant chemoimmunotherapy in locally advanced esophageal squamous cell carcinoma. Cancer Immunol Immunother. 2025 Jun 18;74(8):243. doi: 10.1007/s00262-025-04099-9. PMID 40531216